CLINICAL TRIAL: NCT06825637
Title: The Use of SmartPhone App (Kandoo) to Enhance Efficacy of Brief Behavioral Activation in Reducing Mood Disorder Symptoms
Acronym: Kandoo
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Child Mind Institute (Other)
Collaborators: Fort Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00081465
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Depression Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brief Behavioral Activation with Kandoo (Experimental): Participants will use Kandoo to track their activities while receiving Brief Behavioral Activation treatment.
  Interventions: Device: Kandoo
- Brief Behavioral Activation with traditional paper pencil tracking (No Intervention): Participants will use paper and pencil worksheets to track their activities while receiving Brief Behavioral Activation treatment.

INTERVENTIONS:
Device: Kandoo — Kandoo is an app that allows patients to track their activities in an engaging and gamified platform.
  Arms: Brief Behavioral Activation with Kandoo

SUMMARY:
The current project is a pilot study that seeks to compare the efficacy of Brief Behavioral Activation's treatment-as-usual that uses paper and pencil tools to Kandoo, a digital, gamified version of activity scheduling and self-monitoring, in a diverse sample of youth presenting with clinically significant symptoms of depression. We will compare the level of pre- and post-treatment depressive symptoms in participants, who will participate in an 8-week brief behavioral activation treatment protocol augmented with Kandoo to the pre- and post- treatment depressive symptoms in the control participants, who will participate in 8-week, treatment as usual, brief behavioral activation treatment protocol. To explore treatment response for the clinically significant symptoms, we will obtain pre- and post-treatment measures of depression, global functioning, and patient goals. During the standard clinical intake, additional information will be obtained, including detailed demographics, medical history, mental health status, and social skills. Beyond determining the overall effectiveness of BBA augmented with Kandoo, the sample diversity and availability of clinical behavioral observations of the participants will permit the development of explanatory models of predictive factors for BBA with Kandoo intervention outcomes.

DETAILED DESCRIPTION:
Youth depression is one of the most common psychiatric conditions, affecting 1%-3% of prepubertal children and 3%-9% of adolescents. By late adolescence, between 20-25% of youth will have experienced at least one episode of major depression. Conservative prevalence estimates suggest that in a single year, between 12.5% of 12- to 17-year-olds experience symptoms of a major depressive episode5. Accordingly, pediatric mood disorders, including but not limited to major depressive disorder, are a major public health concern. These issues are serious and potentially lethal. In 15 year follow-up research of children with major depression, 4% died by suicide. In 10- to 15-year follow-up research of adolescents with depression, 8% died by suicide1. Individuals who experience depressive episodes in adolescence are at increased risk for at least one recurrent episode in adulthood. Moreover, youth depression is related to a range of additional poor psychiatric, as well as medical outcomes, such as increased risk of suicidality, higher risk for comorbid psychiatric conditions (e.g., anxiety, substance use, etc.), increased risk of obesity, type 2 diabetes, etc.

Adolescence is a pivotal developmental period that is characterized by the understanding and building of relationships, exploration of interests, development of essential skills needed for adaptive living and professional success, and the transition to higher education and/or the workforce. Depression interferes with these processes and has long-term impact on socioeconomic status, as well as a myriad of psychosocial outcomes: relationship challenges (e.g., familial, peer, romantic, etc.), less perceived social support, lower academic achievement, and attainment, and unemployment2. Even after spontaneous remission or a successful course of treatment, given depressive sequelae (i.e., underdeveloped coping skills, dysfunctional thinking patterns, cognitive distortions, impaired interpersonal relationships, etc.), individuals often require long-term treatment1. Even though treatment for depression is largely effective and untreated depression is associated with more severe prognostic consequences, most individuals with depression do not receive treatment3.

Only about one-third of youth exhibiting clinical psychiatric and behavioral issues access professional care. Low treatment utilization is associated with systematic difficulties (e.g., cost, waitlists, etc.), perceptions towards care providers and the treatment process, issues with the recognition and understanding of psychiatric conditions and related treatment, and characteristics of family systems. Key access to care challenges includes high demands for specialists' services and extensive waitlists5. Decreasing obstacles and increasing facilitators are critical to facilitating youths' access to much needed clinical services. In addition, youth report a range of their own perceptions (e.g., embarrassment, previous experiences, negative expectations, preference to be self-reliant, societal stigma, confidentiality concerns, etc.) as factors that impede their help seeking behaviors and psychiatric health.

Behavioral models of depression maintain that symptoms emerge as an individual has decreased positive experiences and increased negative experiences. As this pattern repeats, activity levels decrease and low mood intensifies, initiating the 'vicious cycle' of depression. Brief Behavioral activation (BBA) has three aims, which are accomplished through activity scheduling and self-monitoring. The first aim is to decrease non-adaptive behaviors, such as avoidance, that maintain depressive symptoms. The second aim is to increase valued, adaptive activities that decrease depressive symptoms. The third aim is problem solving focused on any obstacles and impediments to completing valued adaptive activities. By increasing participation in preferred and rewarding activities, BBA breaks the aforementioned vicious cycle. As participation in preferred and valued activities increases, the individual is reinforced, leading to decreased depressive symptoms. Research demonstrates that BBA is clinically effective at decreasing depressive symptoms in adults and adolescents. The treatment has outcomes consistent with other established depression treatments (e.g., cognitive behavioral therapy, interpersonal therapy, etc.)12.

An essential component of BBA is "homework," which involves participating in an engaging, pleasurable activity, as well as pre- and post-assignment mood tracking. Despite this positive relationship between homework adherence and treatment outcomes, homework completion is consistently low. For youth, although highly variable, completion rates are approximately 50%; this often declines as the treatment sessions progress. Although between session tasks are formulated with the goal of completion, adherence is dependent on the patient's willingness and capacity to independently accomplish the activity. Many factors interfere with independent completion of homework: lack of real time clinician encouragement, live feedback, and support for troubleshooting. Youth report that they value homework and know that it is important for treatment success; however, they concurrently indicate that they do not complete tasks because of low motivation, no interest, lack of support, as well as the perception that the assignments are time consuming. With increased support, such as through an engaging, digital, game-like format, assignment adherence may improve13.

Adolescent mental health is recognized as a highly concerning global health issue. When clinically significant psychiatric symptoms emerge during adolescence, if promptly and effectively treated, the issues are decreased or eliminated prior to adulthood. However, when treatment is not provided, problems persist and/or exacerbate, chronic mental distress is instigated, risk increases for challenges related to academic, professional, economic, social, interpersonal, and adaptive functioning. Efficiently and effectively addressing youth mental health challenges with practical and effective treatments is critically needed. Various initiatives are focused on addressing the increasing prevalence of psychiatric conditions in youth, as well as the challenges associated with accessing effective treatment. The saturation of digital devices and platforms has created opportunities to provide digital therapeutics. As part of its work with the Children and Youth Behavioral Health Initiative (CYBHI), the Child Mind Institute (CMI) has launched an ambitious program to tackle the behavioral health symptoms that impact youth and their families. CMI is strongly focused on improving youth mental health services through the development of next-generation digital therapeutics. CMI has conducted decades of scientific research on pediatric behavioral health challenges based on this work. CMI believes these products have the potential to provide low-cost solutions for conditions such as depression and anxiety. One of the components of the collaboration between CYBHI and CMI is Kandoo, a geolocation-based gaming product intended to help youth develop healthy habits by gamifying components of Brief Behavioral Activation. Although Brief Behavioral Activation is a well-documented, evidence-based, therapeutic avenue, it is still unclear how supplementing the treatment with a digital product will help children and teens in clinical practice. To continue developing Kandoo, CMI wants to better understand the lived experiences of youth, including their existing gaming behaviors.

Significance We have evidence-based treatments for depression, but these are limited by access to services and adherence to the treatments when they can be initiated. By increasing adherence, we can be more efficient in providing services, and the increased efficiency will not only improve outcomes but also save clinician time which can be deployed for the care of more adolescents. Kandoo, a smartphone app, is designed to augment BBA by increasing engagement, adherence, and efficiency of the "homework" component of BBA.

Kandoo may increase treatment efficiency and efficacy for youth with symptoms of adolescent depression. Kandoo uses tablets and smartphones, to digitally deliver the components of brief behavioral activation that are traditionally deployed in a paper/pencil format. Kandoo delivers therapeutic content to individuals in situ (e.g., at school or home) in support of treatment provided directly by clinicians, in-person or remotely. Over the past decade, there has been an explosion of digital mental health products; however, research on the effectiveness of these programs has been limited and less than encouraging. From a resource perspective, supplementing services via a digital app is ideal, as it removes some of the dependencies on the clinic and therapist, as well as resources, such as transportation, which can vary substantially. In addition, it removes the burden of self-monitoring and tracking and, by providing immediately updated information about treatment progress, engaging psychoeducation content, and motivating gamified designs. Digital tools are expected to increase the user's level of treatment engagement and positively impact treatment outcomes. Kandoo was designed to meet these demands, while collecting data on treatment progress and patient status, as well as serving as a screening tool for those who may need additional support.

Gamification has the potential to increase sustained engagement and adherence with interventions. Sustaining engagement is a key challenge for the delivery of treatments, especially when working with depressed youth who are expected to complete homework assignments and otherwise function independently in unstructured or unsupervised settings (e.g., the home). Gamification is a commonly cited means of improving and sustaining engagement, as it can increase motivation through the creation of a positive, reward-driven learning environment that easily and immediately provides feedback3,4. Appealing graphics and other media-based features (e.g., engaging digital psychoeducational content, in-app rewards) are added benefits of gamification; together these features serve to increase motivation for treatment and support and sustain at-home interventions8.

Study Design:

Evaluate the effectiveness of Behavioral Activation, augmented with Kandoo, in a sample of youth with depressive symptoms.

This study will enroll patients receiving BBA from the Child Mind Institute Medical Practice and Forth Health (https://www.forthealth.com/). Fort Health is a virtual mental healthcare service that was built in collaboration with the Child Mind Institute. Fort Health has been designed for children and adolescents, between 4 and 24 years of age. Through online platforms, Fort Health provides accessible, and evidence-based care, including online therapy, parent coaching, and psychiatry services. To ensure coordinated care, therapy, coaching, and psychiatry services are integrated with each other, as well as with the care given by primary care providers. Services are offered in New York, New Jersey, and Pennsylvania, and Illinois and Texas will be added soon. CMI will contract with Fort Health to identify eligible patients in their practice, introduce the study, and conduct BBA therapy. This study will enroll 2 groups:

Group 1 (CMI): This group uses a pre-post-treatment trial design of BBA augmented with Kandoo in 50 youth (males and females, ages 13.0-25.11). We will recruit participants already enrolled in the Child Mind Institute's (CMI) outpatient clinic, which offers treatment to youth with mental health and learning disorders. All participants in this group will receive BBA augmented with Kandoo.

Group 2 (Fort Health): This group uses a control group pre-post-treatment trial design of BBA augmented with Kandoo in 200 youth (males and females, ages 13.0-25.11). CMI will partner with Fort Health to recruit patients for group 2. We will recruit participants already enrolled in Fort Health's Virtual Mental Health clinic, which offers treatment to youth with mental health and learning disorders. Participants in this group will be randomized into either the BBA treatment as usual group (control group) or the BBA augmented with Kandoo group (Kandoo treatment group). One hundred participants will be randomly assigned into each group.

For both groups, clinicians will be informed of the study and will be asked to refer patients who have depressive symptoms and are candidates for BBA therapy. It is expected that the clinical presentation will include depressive symptoms consistent with mild-to-moderate depression. Two of the symptoms are (1) depressed/irritable mood most of the day and (2) markedly diminished interest or pleasure in all, or almost all, activities most of the day, nearly every day.

The standard BBA treatment protocol includes 8 weekly sessions. Study participants and their clinicians are allowed up to 16 weeks to complete the treatment, allowing for typical and expected reasons for missed sessions (e.g., vacation, illness, scheduling difficulties, etc.). Non-study related interventions will be permitted during the course of the study, consistent with standard practice. These situations will be documented. Participants' symptoms will be assessed weekly using the Mood and Feelings Questionnaire (MFQ). Fifty youth will be recruited to the BA + Kandoo Treatment study. The study will use a pre-post study design.

Variables of interest will be measured before, throughout, and at the end of the treatment. A battery of questionnaires examining depression, global functioning, patient goals, in-therapy feedback, and attitudes towards the digital platform will be administered. At sessions 1, 5, and 8, depression, global functioning, and goals measures will be administered. At sessions 2, 3, 4, 6, and 7, the abbreviated depression measure will be administered. In addition, 6 weeks after session 8, the depression measure will be re-administered as extended post-treatment monitoring. Please see Appendix A for a detailed list of the measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 13.0 to 25:11 years old
2. Sex: male and female
3. Currently enrolled as a patient in the CMI clinic or Fort Health Virtual Outpatient Mental Health Clinic
4. Current clinical presentation must include symptoms of mild-to-moderate depression, two of which must be depressed/irritable mood most of the day and markedly diminished interest or pleasure in all, or almost all, activities most of the day, nearly every day
5. Access to a smart device
6. Internet connectivity
7. Approval by parents and clinician for participants 13-17.11; approval by clinician for participants 18+

Exclusion Criteria:

1. Current exclusionary psychiatric conditions are (not others):

   1. eating disorder
   2. manic episode (any current or history)
   3. psychotic episode or psychotic disorder
   4. active suicidality
   5. homicidal
2. Any neurologic impairment that limits the ability to use a touch screen.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptoms and Global Functioning | 8 weeks
  We will compare the pre- and post-treatment depressive symptoms and global functioning of participants, who completed BBA with Kandoo.

SECONDARY OUTCOMES:
Improvement Factors | 8 weeks
  We will explore what factors influenced improved as a result of BBA treatment with Kandoo, including explanatory models of predictive factors for BBA with Kandoo intervention outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milham, MD, PhD, Principal Investigator — Child Mind Institute
Locations (1):
- Child Mind Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No